CLINICAL TRIAL: NCT02886611
Title: Limbal Stem Cell Deficiency of Genetic Origin: Genotype-phenotype Correlation
Acronym: SILOG
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: EGN_2015_36
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Limbus Corneae

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
The study aims at searching for a genotype-phenotype correlation in patients with a genetic pathology of the ocular surface, in order to identify genetic abnormalities associated with the most severe clinical situations.

ELIGIBILITY:
Inclusion Criteria:

* genetic pathology of ocular surface

Exclusion Criteria:

* Agonal glaucoma
* Low vision mostly related to retinal pathology
* Pregnant or breast feeding patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with decreased visual acuity of corneal origin will be selected and genetic analysis will be performed.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-12-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Genotype-phenotype Correlation | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Anna GEMAHLING, MD, Principal Investigator — Hôpital Fondation Adolphe de Rothschild; Eric GABISON, MD, Principal Investigator — Hôpital Bichat (AP-HP); Dominique BREMOND-GIGNAC, MD, Principal Investigator — Hopital Necker-enfants malades (AP-HP)
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France